CLINICAL TRIAL: NCT04420793
Title: Voice Analysis in Patients Receiving Electroconvulsive Therapy
Brief Title: Voice Changes During ECT
Acronym: VAPRE
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 00089198
Record Dates: First submitted 2020-03-10; First posted 2020-06-09 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Unipolar Depression; Bipolar Depression; Bipolar Disorder, Manic
Keywords: VAPRE
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ECT and Voice Recorded Group: This is an add-on study of voice samples to be gathered during ECT clinical treatments. The ONLY research procedures are four tasks on an online form, one text task and three voice recording tasks. These voice recordings will take place in a private room on the 5th floor of the Institute of Psychiatry on the same day of a patient's ECT treatment. The questionnaire will take less than 10 minutes.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — 3 voice recording tasks and 1 text entry task will be performed.

SUMMARY:
Depressed patients talk differently when they are depressed compared to when they are well. But it is hard to actually measure what the differences are. The study team will record voice samples from patients with mood disturbances, like depression, over the course of their receiving an electroconvulsive therapy (ECT) series. The study team will try and measure or quantify exactly what has changed in their speech and voice. The study team will choose ECT as it is one of the most effective and rapid treatment for depression. The study team will use a service provided by a company, NeuroLex, who has complex computer programs (artificial intelligence, AI) to analyze the voice samples.

ELIGIBILITY:
INCLUSION CRITERIA:

* Any candidate for electroconvulsive therapy who is about to initiate their ECT course at Medical University of South Carolina (MUSC) for a clinically indicated diagnosis
* Age 18 to 90 years old
* Able to speak and understand English
* Able to give consent to participate in the study

EXCLUSION CRITERIA:

* Any medical condition that limits the ability to speak or speak clearly, for example a history of head and/or neck cancer, spinal cord injury affecting speech, amyotrophic lateral sclerosis, or those with absence of critical anatomical structures involved in speech.
* Any voice characteristics that may limit the ability to speak English clearly including speech impediments or heavy accents (as evidenced by the pronunciation of the English language in such a non-standard way that research staff). If study staff have significant difficulty understanding the participant's responses in conversation, this may warrant exclusion.
* Patients who are receiving ECT by involuntary order, by order of their guardian, or by a court order, as evidenced by patient report or brief chart review.
* Patients who elect to not receive their full course of ECT at MUSC.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing electroconvulsive therapy (ECT) at the Medical University of South Carolina on an outpatient or inpatient basis.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Acoustic feature: zero crossing rate | Throughout a course of electroconvulsive therapy (ECT) which may last between 2 and 7 weeks.
  crossings per second
Acoustic feature: energy and entropy | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  decibels
Acoustic feature: spectral centroid, spectral spread, spectral entropy, spectral flux, spectral rolloff | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  hertz
Acoustic feature: Mel-Frequency Cepstral Coefficients, Chroma Vectors, and Chroma Deviation | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  unitless
Linguistic features: question ratio, filler ratio, number ratio, type token ratio | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  unitless ratio
Linguistic features: verb frequency, noun frequency, pronoun frequency, adverb frequency, adjective frequency, particle frequency, conjunction frequency, pronoun frequency | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  percentage
Linguistic features: standardized word entropy | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  decibels/log(total word count)
Linguistic features: Brunets index | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  W (lexical richness)
Linguistic features: Honores statistic | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  R (lexical richness)
Linguistic features: rate of speech | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  words per minute
Meta-features: fatigue | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Machine learning approach to evaluate binary outcome: fatigued or awake
Meta-features: audio quality | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Machine learning approach to evaluate binary outcome: bad or good
Meta-features: sentiment | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Machine learning approach to evaluate binary outcome: sad or happy
Meta-features: stress | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Machine learning approach to evaluate binary outcome: stressed or not stressed
Meta-features: gender | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Machine learning approach to evaluate binary outcome: male or female
Meta-features: accent | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Machine learning approach to evaluate a categorical outcome of accent region: england, indian, australian, etc.
Meta-features: length | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  seconds
Meta-features: age | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Machine learning approach to evaluate estimated decade-age: 10s, 20s, 30s, 40s, 50s, 60s, 70s, 80s, 90s, etc.
Comparing the voice feature(s) with greatest statistically significant change to Patient Health Questionnaire (PHQ)-9 scores | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  The voice feature(s) found to have changed most significantly will be compared to Patient Health Questionnaire-9 scores which approach a total score that is less than 8, indicative of reduced depressive symptoms throughout Electroconvulsive Therapy
Acoustic Feature Specific Changes within and across sessions | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Generalized mixed linear model will be used to evaluate which acoustic features change with P value threshold of <0.05
Linguistic Feature Specific Changes within and across sessions | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Generalized mixed linear model will be used to evaluate which linguistic features change with P value threshold of <0.05
Meta-Feature Specific Changes within and across sessions | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Generalized mixed linear model will be used to evaluate which meta features change with P value threshold of <0.05

SECONDARY OUTCOMES:
Acoustic Feature Specific Changes between sessions | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Acoustic voice features will be evaluated using continuous averages using one sample t-tests and we will be testing the difference over time to a null hypothesis of 0 (for no change) in the one sample t-test.
Linguistic Feature Specific Changes between sessions | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Linguistic voice features will be evaluated using continuous averages using one sample t-tests and we will be testing the difference over time to a null hypothesis of 0 (for no change) in the one sample t-test.
Meta-Feature Specific Changes between sessions | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Meta-voice features will be evaluated using continuous averages using one sample t-tests and we will be testing the difference over time to a null hypothesis of 0 (for no change) in the one sample t-test.
Patient Chart Review Data: Age | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  years
Patient Chart Review Data: inpatient/outpatient status | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  binary: inpatient or outpatient
Patient Chart Review Data: gender | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  male, female, unspecified
Patient Chart Review Data: race | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  african american, caucasian, hispanic, asian american, etc.
Patient Chart Review Data: Psychiatric diagnosis for ECT | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Diagnosis indicated for receiving ECT
Patient Chart Review Data: PHQ-9 score at each session | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Total (0-27) on 9 question scale
Patient Chart Review Data: Psychiatric hospitalizations | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Number
Patient Chart Review Data: Past Psychiatric Medication Trials | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Number
Patient Chart Review Data: Current Psychiatric Medication Trials | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Number
Patient Chart Review Data: Classes of Current Psychiatric Medications | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Categorical: Sedative, Selective Serotonin Reuptake Inhibitor, etc.
Patient Chart Review Data: Suicidal Ideation at ECT consult | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Binary: yes/no
Patient Chart Review Data: Past Suicide Attempts | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Number
Patient Chart Review Data: Psychiatric Review of Systems | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Descriptive, categorical
Patient Chart Review Data: Family Psychiatric History | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Categorical regarding psychiatric diagnoses of family members
Patient Chart Review Data: Number of non-psychiatric medical diagnoses | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Number
Patient Chart Review Data: Past non-psychiatric medication trials | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Number
Patient Chart Review Data: Current non-psychiatric Medications | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Number
Patient Chart Review Data: Tobacco use history | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Binary (yes/no)
Patient Chart Review Data: Tobacco use pack year | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  pack-year (total years smoked*average packs per day)
Patient Chart Review Data: Prior ECT treatment | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Binary (yes/no)
Patient Chart Review Data: total # of prior ECT treatments for response in the past | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Numerical
Patient Chart Review Data: Prior transcranial magnetic stimulation (TMS) treatment | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Binary (yes/no)
Patient Chart Review Data: Prior response to ECT or TMS | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Categorical
Patient Chart Review Data against voice features | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  We will evaluate voice features with statistically significant changes against respective participant chart review data using a general linear model with a clustering component for repeated measures which may also be applied to contrast statements evaluating overall change over time (from baseline to end).
Generating ROC curves: stress | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Clinically determined stress level (mood) will be compared to meta-feature extractions of stressed vs. not stressed from voice recordings will be used to calculate an area under the receiver operating curve (AUOC)
Generating ROC curves: fatigue | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Clinically determined fatigue (motor) will be compared to meta-feature extractions of fatigued vs. awake from voice recordings will be used to calculate an area under the receiver operating curve (AUOC)
Generating ROC curves: sentiment | Throughout a course of electroconvulsive therapy which may last between 2 and 7 weeks.
  Clinically determined sentiment (affect and mood) will be compared to meta-feature extractions of happy vs. sad from voice recordings will be used to calculate an area under the receiver operating curve (AUOC)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Christensen, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No